CLINICAL TRIAL: NCT06434467
Title: The Efficacy and Safety of Nelarabine Injection in the Treatment of Refractory or Recurrent T-lymphoblastic Leukemia (T-ALL) and T-lymphoblastic Lymphoma (T-LBL) in Children and Adults
Brief Title: The Efficacy and Safety of Nelarabine Injection in Patients With T-lymphoblastic Leukemia and T-lymphoblastic Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLB-III-01
Record Dates: First submitted 2024-05-17; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-11

CONDITIONS: T-lymphoblastic Leukemia; T-lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — nelarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nelarabine injection (Experimental): Adults (≥18 years old): 1500 mg/m², administer intravenously for at least 2 hours on days 1, 3, and 5, repeating every 21 days.
  Children (1-17 years old): 650 mg/m ², administer intravenously for 1 hour daily for 5 consecutive days, repeating every 21 days.
  Interventions: Drug: Nelarabine injection

INTERVENTIONS:
Drug: Nelarabine injection — Nelarabine is a prodrug of the nucleotide metabolism inhibitor deoxyguanosine analogue 9-β-arabinoguanine (ARA-G). Nelarabine undergoes catalytic transformation by adenosine deaminase (ADA), resulting in the removal of its methoxy group and conversion into ARA-G, Subsequently, ARA-G undergoes sequential monophosphorylation by deoxyguanosine kinase and deoxycytosine nucleoside kinase, yielding the active compound 5'-Guanosine triphosphate (GTP), ARA-GTP. This active compound accumulates within leukemic blast cells and binds to deoxyribonucleic acid (DNA), effectively inhibiting DNA synthesis and ultimately leading to cell death.

SUMMARY:
This is a single-arm, open-label, multicenter, phase III clinical study that aims to evaluate the efficacy and safety of Nelarabine injection in the treatment of refractory or recurrent T-lymphoblastic leukemia (T-ALL) and T-lymphoblastic lymphoma (T-LBL) in both children and adults. The trial includes 83 subjects, consisting of 35 adults and 48 children, and aims to evaluate the composite complete response rate (CCR) within 2 cycles, assessed by the Independent Review Committee (IRC), following treatment with Nelarabine injection for children and adults with refractory or recurrent T-ALL and T-LBL.

The sample size of this study is estimated according to the treatment period of 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined this study, signed an informed consent form, and had good compliance;
* Age: ≥ 1 year old and ≤ 65 years old (if the child has no reading ability, the child's immediate family/guardian can fully read the informed consent form, sign and witness the informed consent process); Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0-2 points; Expected survival period exceeds 3 months;
* Subject population:

  1. According to the revised classification criteria for myeloid tumors and acute leukemia in 2016, morphology, immunology, cytogenetic and molecular (MICM) classification and/or pathological and imaging diagnosis confirmed by local laboratories as T-ALL or T-LBL stage II-IV;
  2. Philadelphia chromosome negative (Ph -);
  3. Difficult to treat or disease recurrence status;
  4. Previously received two chemotherapy regimens without response, or experienced recurrence after treatment.
* The main organ functions well and meets the following standards:

  1. Biochemical examination must meet the following standards:

     Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN) (if T-ALL/T-LBL affects the liver, total bilirubin ≤ 3 times the upper limit of normal value); Alanine transferase (ALT) and aspartate transferase (AST) ≤ 3 × ULN (if T-ALL/T-LBL affects the liver, ALT and/or AST ≤ 5 × ULN);

     Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate estimated based on Cockcroft Gault glomerular filtration formula ≥ 50 mL/min.
  2. The coagulation function test needs to meet the following standards: prothrombin time (PT), activated partial thromboplastin time (APTT), international standardized ratio (INR) ≤ 1.5 x ULN (without receiving anticoagulant treatment).
* Before starting to use the investigational drug, all non hematological toxicity (except for hair loss and fatigue) of previous anti leukemia treatments must have been restored to level 1 or baseline levels ((NCI Common Terminology Criteria for Adverse Events(CTCAE) version5.0));
* Female participants of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 6 months after the end of the study; Within 7 days prior to enrollment, the serum pregnancy test was negative and must be a non lactating subject; Male participants should agree to adopt avoidance measures during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Previous treatment:

  1. Within 3 weeks prior to the first medication, chemotherapy (including intrathecal injection, excluding ALL/LBL maintenance therapy) was received. Within 12 weeks prior to the first medication, radiation therapy (brain spine, pelvis, and other radiation areas exceeding 25% of the total bone marrow volume), immune checkpoint inhibitors, Chimeric Antigen Receptor T-Cell (CAR-T) Therapy were received. Other small molecule anti-tumor treatments received before the first medication (washout period calculated from the end of the last treatment) were within 5 half-lives;
  2. Within 7 days prior to the first administration, receive ≥ 5 days of intravenous or oral prednisone ≥ 30mg/m2 or an equal amount of other glucocorticoids. Within 28 days prior to the first administration, receive ≥ 14 days of intravenous or oral prednisone ≥ 30mg/m2 or an equal amount of other glucocorticoids. Single dose prevention or treatment of airway stenosis is allowed to be used; Note: If the patient's white blood cell (WBC) is ≥ 30 × 10^9/L, or if the liver, spleen, or lymph nodes are significantly enlarged; Patients with tumor lysis characteristics (biochemical tests, etc.) may undergo pre-treatment, and the use of prednisone/dexamethasone ± cyclophosphamide during the pre-treatment period is allowed to prevent tumor lysis syndrome;
  3. Vaccination received within 4 weeks prior to the first medication, or planned vaccination during the study period;
  4. Participated in clinical trials of other anti-tumor drugs within 4 weeks prior to the first medication use;
  5. According to the researcher's judgment, there are individuals with accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study, or individuals who are deemed unsuitable for enrollment due to other reasons.
* Concomitant diseases and medical history:

  1. Has experienced or currently suffers from other malignant tumors within 3 years prior to the first medication use. The following two situations can be included in the study: achieving disease-free survival (DFS) for 5 consecutive years for other malignant tumors treated with a single surgery; Cured cervical cancer in situ, thyroid cancer, non melanoma skin cancer, and superficial bladder tumors [Ta (non invasive tumor), Ti (carcinoma in situ), and T1 (tumor infiltrating basement membrane)];
  2. Unresolved neurotoxicity of ≥ CTC AE II grade due to any previous treatment;
  3. Within 28 days prior to the start of the research treatment, significant surgical treatment, open biopsy, and obvious traumatic injury were received;
  4. Within 3 months prior to the first medication, there have been incidents of arterial/venous thrombosis, such as cerebrovascular accidents (including cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
  5. Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
  6. Within 6 months prior to the first medication, the patient had ≥ grade 2 myocardial ischemia or infarction, arrhythmia (QTcF>450ms in males and>470ms in females), ≥ grade 2 congestive heart failure (NYHA classification), and left ventricular ejection fraction (LVEF) assessed by echocardiography<50%.
  7. Existence of active infection (≥ CTC AE level 2 infection);
  8. Active hepatitis *; Hepatitis B reference: hepatitis B virus (HBV) DNA detection value ≥ upper limit of normal value; Hepatitis C reference: hepatitis C virus (HCV) antibody positive, and HCV virus titer detection value exceeds the upper limit of normal value;
  9. Individuals with a history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
  10. Have a history of epilepsy;
  11. Have a history of Down syndrome;
  12. Merge central nervous system leukemia/lymphoma.
* The patient plans to receive chest radiation therapy.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Composite complete response rate (CCR) assessed by the Independent Review Committee (IRC) | During the study period (Baseline up to two months)
  Proportion of complete responses (CCR) after 2 cycles of antineoplastic therapy as determined by independent review committee (IRC) assessment

SECONDARY OUTCOMES:
Composite complete response rate (CCR) assessed by the investigator | During the study period (Baseline up to two months)
  Proportion of complete responses (CCR) after 2 cycles of antineoplastic therapy as determined by the investigator.
Objective Remission Rate (ORR) | During the study period (Baseline up to two months)
  The best Objective Remission Rate (ORR) for both complete response (CR) and partial response (PR) cases within 2 cycles.
Duration of complete remission (DOCR) | During the study period (Baseline up to two years)
  Proportion of patients whose tumor shrinks or stabilizes for some time, including cases of complete response (CR), partial response (PR), and stable disease (SD).
Disease-free survival (DFS) | During the study period (Baseline up to two years)
  It refers to the time from the first day of absence of disease to the recurrence of disease.
Overall survival (OS) | During the study period (Baseline up to two years)
  It indicates the time interval from randomization to death from any cause.
Incidence of adverse events (AEs) | During the study period (Baseline up to two years)
  Adverse events refer to all adverse medical events that occur after a patient or clinical trial subject receives an experimental drug, which can be expressed as symptoms, signs, diseases, or abnormalities in laboratory tests, but are not necessarily related to the treatment of the experimental drug.
Incidence of serious adverse events (SAEs) | During the study period (Baseline up to two years)
  Serious adverse events include death, life-threatening, permanent or serious disability or loss of function, hospitalization or prolonged hospitalization, and adverse medical conditions such as congenital abnormalities or birth defects.
Peak time (Tmax) | During the study period (Baseline up to two years)
  Time to maximum plasma concentration.
Peak concentration(Cmax) | During the study period (Baseline up to two years)
  Pharmacokinetic parameters, including but not limited to: Peak concentration(Cmax)
Half-life(t1/2) | During the study period (Baseline up to two years)
  It is the time required for half of the drug to be eliminated from the plasma
Negative rate of minimal residual disease in bone marrow (MRD) | During the study period （Baseline up to two years)
  The proportion of trace leukemic cells negative in patients with hematologic tumors after treatment.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Aerospace Medical Center, Beijing, Beijing Municipality
  - Beijing Tongren Hospital,CMU, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Army Military Medical University, Chongqing, Chongqing Municipality
  - The first hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Prevention Center, Guangzhou, Guangdong
  - Cancer Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Yulin Red Cross Hospital, Yulin, Guangxi
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Affiliated cancer hospital of harbin medical university, Harbin, Heilongjiang
  - Institute of Hematology & Oncology, Harbin First Hospital, Harbin, Heilongjiang
  - Henan Children's Hospital, Zhengzhou, Henan
  - Tongji Medical College of HUST, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Nanjing childrens Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The First Hospital Of Jilin University, Changchun, Jilin
  - Weihai Municipal Hospital, Weihai, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - Sichuan Academy of Medical Sciences · Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang